CLINICAL TRIAL: NCT06526780
Title: Bronchoscopy Versus Imaging in Diagnosis of Airway Diseases in Critically Ill Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AA Nagy, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BVIAD
Record Dates: First submitted 2024-07-19; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Airway Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Critical ill children with airway diseases
  Interventions: Procedure: Bronchscopy

INTERVENTIONS:
Procedure: Bronchscopy — Bronchscopy in critical ill children with airway diseases
  Other Names: chest computed tomography scan with virtual bronchscopy

SUMMARY:
Patients with suspected airway illness often go through a diagnostic assessment that includes chest radiographs, Computed tomography scans, and fiber optic bronchoscopy.

DETAILED DESCRIPTION:
A correct diagnosis is necessary for effective therapy of airway illness. Usually necessary for these invasive treatments. The "gold standard" for tracheobronchial pathology identification and diagnosis is rigid or fiber optic bronchoscopy. Fiber Optic is a procedure that is generally safe, although it can have negative effects, particularly in patients who are at greater risk. Therefore, it is important to continually develop and improve non-invasive procedures that enable airway examination.

The laryngotracheal and bronchial airway is affected by a wide range of diseases, and imaging is essential for assessing these anomalies. The location, scope, and type of these lesions may be determined with great accuracy using computed tomography.

Bronchoscopy allows direct visualization of trachea and bronchi by rigid open tube bronchoscope or flexible fiber optic scope. Detailed evaluation of airways with bronchoscopy offers advantages over other diagnostic tools and allows interventional procedures such as biopsy of lesions, removal of foreign bodies, dilatations of stenosis and obtaining samples for cytological and microbiologic analysis.

Bronchoscopy can be performed either by rigid or flexible instruments depending on the needs of patients. The pediatric airway is notably different from adults. It is smaller in size, larynx and tracheal proportion is more as compared to adults and epiglottis is more posterior and narrower .

Fiber Optic bronchoscopy with or without bronchoalveolar lavage is particularly important in the diagnosis and treatment of specific respiratory problems in critically ill infants and children hospitalized in the pediatric Intensive care unit.These comprise situations such as segmental lung collapse, pulmonary infections including community-acquired and ventilator-associated pneumonia, pulmonary infections in immunocompromised hosts, and pulmonary bleeding. In addition, bronchscopy has a special role in airway problems in very sick pediatric patients. It may be crucial in intubation of the difficult airways and in the assessment of airway anomalies.

There are various indications for bronchoscopy: persistent stridor , congenital, anatomical, or acquired anomalies, persistent wheezing, hemoptysis, persistent or recurring atelectasis, persistent or recurring pneumonia, and localized hyperinflation. Other uses of bronchoscopy are bronchoalveolar lavage , getting biopsy samples, and aspiration of secretions. Examples of therapeutic bronchoscopy are administering medications and removing foreign bodies.

Absolute contraindications for bronchoscopy include severe hypoxemia, hemodynamic instability, and uncorrected hemorrhagic diathesis. Severe pulmonary hypertension and congenital cyanotic cardiomyopathy with increased bronchial collateral circulation are relative contraindications. In addition, instabilities in the cervical spine or atlanto occipital transition are considered relative contraindications for rigid bronchoscopy.

The common complication of bronchoscopy is related to anesthesia, mechanical trauma ( epistaxis , pneumothorax, and hemoptysis), hypoxemia, laryngospasm, post-lavage fever, and infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 month: 18 years.
* Critically ill patients with suspected airway diseases for the following indications:
* Difficult intubation.
* extubation failure (defined as the replacement of an endotracheal tube within <48 h after extubation).
* Persistent stridor. •Acute unexplained respiratory distress.• Localized hyperinflation.
* Suspected foreign body.
* Persistent and recurrent wheezes.
* Persistent and recurrent atelectasis.
* Unexplained hemoptysis

Exclusion Criteria:

* Age ( < 1month and > 18 years )
* Severe hypoxemia
* Hemodynamic instability
* Uncorrected bleeding diathesis
* Unresolved lung infection

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Visualization of airway abnormalities by bronchscopy | During procedure
  Direct visualization of airway by bronchscopy
Visualization of airway abnormalities by computed tomography scan | During procedure
  Assessment of airway by computed tomography scan with virtual bronchscopy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Midulla F, de Blic J, Barbato A, Bush A, Eber E, Kotecha S, Haxby E, Moretti C, Pohunek P, Ratjen F; ERS Task Force. Flexible endoscopy of paediatric airways. Eur Respir J. 2003 Oct;22(4):698-708. doi: 10.1183/09031936.02.00113202. PMID 14582925
- [Result] Sinha V, Gurnani D, Barot DA. A study of applications of rigid bronchoscopy in pediatric patients. Indian J Otolaryngol Head Neck Surg. 2014 Jun;66(2):142-4. doi: 10.1007/s12070-013-0667-1. Epub 2013 Jun 27. PMID 24822151
- [Result] Wood RE. Evaluation of the upper airway in children. Curr Opin Pediatr. 2008 Jun;20(3):266-71. doi: 10.1097/MOP.0b013e3282ff631e. PMID 18475094
- [Result] Davidson MG, Coutts J, Bell G. Flexible bronchoscopy in pediatric intensive care. Pediatr Pulmonol. 2008 Dec;43(12):1188-92. doi: 10.1002/ppul.20910. PMID 19009620
- [Result] Soong WJ, Shiao AS, Jeng MJ, Lee YS, Tsao PC, Yang CF, Soong YH. Comparison between rigid and flexible laser supraglottoplasty in the treatment of severe laryngomalacia in infants. Int J Pediatr Otorhinolaryngol. 2011 Jun;75(6):824-9. doi: 10.1016/j.ijporl.2011.03.016. Epub 2011 Apr 21. PMID 21513991
- [Result] Levin R, Kissoon N, Froese N. Fibreoptic and videoscopic indirect intubation techniques for intubation in children. Pediatr Emerg Care. 2009 Jul;25(7):473-9; quiz 480-2. doi: 10.1097/PEC.0b013e3181aba8c1. PMID 19606008
- [Result] Faro A, Wood RE, Schechter MS, Leong AB, Wittkugel E, Abode K, Chmiel JF, Daines C, Davis S, Eber E, Huddleston C, Kilbaugh T, Kurland G, Midulla F, Molter D, Montgomery GS, Retsch-Bogart G, Rutter MJ, Visner G, Walczak SA, Ferkol TW, Michelson PH; American Thoracic Society Ad Hoc Committee on Flexible Airway Endoscopy in Children. Official American Thoracic Society technical standards: flexible airway endoscopy in children. Am J Respir Crit Care Med. 2015 May 1;191(9):1066-80. doi: 10.1164/rccm.201503-0474ST. PMID 25932763
- [Result] Schramm D, Freitag N, Nicolai T, Wiemers A, Hinrichs B, Amrhein P, DiDio D, Eich C, Landsleitner B, Eber E, Hammer J; Special Interest Group on Pediatric Bronchoscopy of the Society for Pediatric Pneumology (GPP) and invited Societies involved in pediatric airway endoscopy. Pediatric Airway Endoscopy: Recommendations of the Society for Pediatric Pneumology. Respiration. 2021;100(11):1128-1145. doi: 10.1159/000517125. Epub 2021 Jun 7. PMID 34098560
- [Result] Rosenthal M. Bronchoscopy and infection. Paediatr Respir Rev. 2003 Jun;4(2):143-6. doi: 10.1016/s1526-0542(03)00025-3. PMID 12758052